CLINICAL TRIAL: NCT06271473
Title: Comparative Study Between Pars Plana Vitrectomy With Internal Limiting Membrane Peeling With or Without Planned Foveal Detachment for Management of Non-tractional Refractory Diabetic Macular Edema
Brief Title: Effect of PPV+ILM Peeling +/- Subretinal Injection of Ringer Lactate in Management of Nontractional Refractory DME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AinShamsU3
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-02

CONDITIONS: Efficacy; Safety
Keywords: refractory diabetic macular edema; internal limiting membrane peeling; pars plana vitrectomy; subretinal injection of ringer lactate
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Intervention Model Description: 20 eyes of 20 patients will be divided randomly into 2 groups:
  * Group (A): 10 eyes subjecting to vitrectomy + ILM peeling only
  * Group (B): 10 eyes subjecting to vitrectomy + ILM peeling + planned foveal detachment via subretinal injection of ringer's solution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjecting to vitrectomy + ILM peeling only (Active Comparator)
  Interventions: Procedure: vitrectomy + ILM peeling +/- planned foveal detachment via subretinal injection of ringer's solution.
- subjecting to vitrectomy + ILM peeling + planned foveal detachment (Active Comparator)
  Interventions: Procedure: vitrectomy + ILM peeling +/- planned foveal detachment via subretinal injection of ringer's solution.

INTERVENTIONS:
Procedure: vitrectomy + ILM peeling +/- planned foveal detachment via subretinal injection of ringer's solution. — vitrectomy + ILM peeling +/- planned foveal detachment via subretinal injection of ringer's solution.

SUMMARY:
To evaluate the efficacy and safety of combined pars plana vitrectomy and planned foveal detachment through subretinal injection of ringer's solution in patients with non-tractional refractory diabetic macular edema.

DETAILED DESCRIPTION:
In non-tractional cases, PPV allows a more efficient clearance of VEGF and other cytokines from the retina and improves retinal oxygenation by promotion of intraocular fluid currents, and relief of any subclinical tractional forces, thereby reducing DME.

To evaluate the efficacy and safety of combined pars plana vitrectomy and planned foveal detachment through subretinal injection of ringer's solution in patients with non-tractional refractory diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Age: above 40 years old.

  * Patients with type two diabetes mellitus of more than 5 years duration.
  * Patients with Best corrected visual acuity better than 3/60.
  * Central macular thickness (CMT) of more than 250 μm despite undergoing six monthly injection of anti-VEGF therapy or corticosteroid or less than 10% reduction in CMT at the last follow up visit.
  * No evidence of vitreomacular traction.
  * Lens status: Pseudophakia or clear crystalline lens.

Exclusion Criteria:

Other causes of macular edema (intraocular inflammation, retinal vein occlusion, Irvin-gass syndrome, pharmacological).

* Ischemic maculopathy by FFA.
* Presence of bad prognostic signs in OCT such as disorganization of inner retinal layers (DRIL) and extensive disruption of IS-OS junction subfoveally.
* Presence of apparent retinal pigment epithelium (RPE) atrophy at or near the macula.
* Presence of proliferative diabetic fibrovascular membranes threatening or at the macula.
* Presence of diabetic optic atrophy or neuropathy.
* Presence of neovascular glaucoma.
* Cataractous lens either preoperatively or as intra or postoperative complication.
* Vitrectomized Eyes.
* A prior intraocular surgery within the past six-months.
* Lost follow up

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
change in CMT by OCT at final visit | after 1 month and 3 months
  decrease or increase in central macular thickness by OCT

SECONDARY OUTCOMES:
change in BCVA at final visit | after 1 month and 3 months
  decrease or increase in best corrected visual acuity

OTHER OUTCOMES:
any surgical complication or recurrence of DME | after 1 month and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman G Salman, MD, Principal Investigator — professor at Ain Shams university
Locations (1):
- Ain Shams university, Cairo, Egypt